CLINICAL TRIAL: NCT05560607
Title: An Open-label, Non-randomized, Multiple-dose Study to Assess the Knockdown of Hepatic HSD17B13 mRNA Expression, Pharmacokinetics, Safety, and Tolerability Following Administration of AZD7503 in Participants With Non-alcoholic Fatty Liver Disease
Brief Title: Knockdown of HSD17B13 mRNA, Pharmacokinetics, Safety, and Tolerability, of AZD7503 in Non-Alcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D9230C00003
Record Dates: First submitted 2022-08-09; First posted 2022-09-29 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Non-alcoholic Fatty Liver Disease; Fatty Liver, Nonalcoholic; NAFLD; Nonalcoholic Fatty Liver Disease; Nonalcoholic Steatohepatitis; NASH
Keywords: NASH; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intervention/ Drug (Experimental): Investigation of the knockdown of hepatic HSD17B13 mRNA expression, PK, safety, and tolerability following multiple dose administration of AZD7503 in male participants and female participants of non-childbearing potential with NAFLD or NASH
  Interventions: Drug: AZD7503 Intervention

INTERVENTIONS:
Drug: AZD7503 Intervention — Part A: Participants will be screened for histologic evidence of NAFLD or NASH and all eligibility criteria in part A prior to enrollment in part B.
  Part B: Participants consented to part B will be administered the study drug over the course of 31 days. At the end of the study a liver biopsy will be collected to measure for endpoints.

SUMMARY:
This is a two-part study. In Part A, eligible participants will undergo a baseline diagnostic liver biopsy to determine non-alcoholic fatty liver disease (NAFLD) Activity Score (NAS) and fibrosis stage, but will not receive study intervention. In Part B, participants with histologically confirmed NAFLD or non-alcoholic steatohepatitis (NASH) will receive study intervention.

DETAILED DESCRIPTION:
This is a single center, open-label Phase I study to assess knockdown of hepatic HSD17B13 mRNA pharmacokinetics (PK), safety, and tolerability following multiple doses of AZD7503 in male and/or female participants of non-childbearing status with NAFLD or NASH.

In Part A, participants at high risk for NAFLD/NASH meeting inclusion criteria for Part A (Section 5.1) and none of the exclusion criteria noted in Section 5.2 will undergo a diagnostic, baseline liver biopsy per standard clinical care. Participants will be consented for the liver biopsy as a first step to determine eligibility for Part B. In Part B, participants will be consented for study intervention administration and repeat liver biopsy at the end-of-treatment (EOT). Eligible participants will be assigned to 1 study intervention cohort. Two additional cohorts may be added based on data from the FiH study (D9230C00001) and emerging data from this study.

Participants who are selected for Part B based on histopathology evaluation (NAFLD or NASH with NAS of ≥3) will have an assessment of the hepatic HSD17B13 mRNA expression from both the liver biopsy obtained in Part A and the liver biopsy obtained at the end of study intervention administration in Part B. The assessments for hepatic HSD17B13 mRNA expression will be performed after each dose cohort is treated and before moving to the next dose cohort.

ELIGIBILITY:
Inclusion Criteria # Part A

1. Participant must be ≥ 18 to ≤ 70 years of age at the time of signing the informed consent.
2. Participants with suspected or confirmed NAFLD or NASH including laboratory values with any of the following deviations at screening

   1. ALT > ULN,
   2. Imaging demonstrating hepatic steatosis including controlled attenuation parameter (CAP) >290 dB/m, OR Liver stiffness of >7.1 kPa as measured by Fibroscan.
3. Body mass index (BMI) ≥20 kg/m2.
4. Male and /or female of non-child bearing potential.

   Inclusion Criteria # Part B
5. Histologic evidence of NAFLD or NASH with a NAS ≥3 following baseline liver biopsy.

Exclusion Criteria:

1. History or presence of hepatic disease (with the exception of hepatic steatosis, NASH) or evidence of other known forms of known chronic liver
2. History of liver transplant, evidence of cirrhosis, or current placement on a liver transplant
3. Positive results for HIV antigen and hepatitis B surface antigen If a participant has a positive result at the screening visit for hepatitis C antibody, the investigator will document that the participant has hepatitis C RNA below the limit of detection and has not received curative treatment in the last 3 years.
4. History of alcohol abuse or excessive intake of alcohol as judged by the investigator.
5. Uncontrolled blood pressure, defined as any of the following during pre-screening and/or Day -1 (mean of 3 measurements):

   1. Systolic blood pressure >160 mmHg.
   2. Diastolic blood pressure >100 mmHg.
6. Any clinically important abnormalities in rhythm, conduction or morphology of the resting ECG.
7. Any clinically important abnormalities in clinical chemistry, hematology, or urinalysis results,
8. Known or suspected history of drug abuse as judged by the investigator.
9. Positive screen for drugs of abuse at screening or admission to the study site prior to the administration of the study intervention.
10. Changes to any concomitant medication (initiation, dose change, or cessation) within one month prior to the screening visit.
11. Any laboratory values with following deviations at screening (one re-test allowed):

    1. (a) ALT >3X ULN
    2. (b) AST >3X ULN
    3. (c) TBL >ULN or INR ≥1.3
    4. (d) ALP >1.5X ULN
    5. (e) eGFR <60 mL/min/1.73 m2 (calculated using CKD Epidemiology Collaboration
    6. [CKD-EPI] formula) and applying the standard correction factor for African
    7. American to the (CKD-EPI) by multiplying the GFR estimate by 1.159 and
    8. confirmed.
    9. (f) Platelets <150 × 109/L

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs). | 99 days
  To assess adverse events as a variable of safety and tolerability of AZD7503.

SECONDARY OUTCOMES:
Change in HSD17B13 mRNA Expression | 31 days
  HSD17B13 mRNA expression from baseline to Day 31 will be assessed
Number of participants with positive anti-drug antibodies to AZD7503 | 99 days
  To explore the formation of ADAs.
Area under plasma concentration time-curve from zero to infinity (AUCinf) of AZD7503 | 99 days
  To characterise the PK (AUCinf) of AZD7503 following SC administration of AZD7503
Area under the plasma concentration-curve from zero to the last quantifiable concentration (AUClast) of AZD7503 | 99 days
  To characterize the PK (AUClast) of AZD7503 following SC administration of AZD7503.
Maximum observed plasma (peak) drug concentration (Cmax) of AZD7503 | 99 days
  To characterise the PK (Cmax) of AZD7503 following SC administration of AZD7503.
Time to reach peak or maximum observed concentration or responsefollowing drug administration (tmax) of AZD7503 | 99 days
  To characterise the PK (tmax) of AZD7503 following SC administration of AZD7503.
Half-life associated with terminal slope (λz) of a semi logarithmic concentration time curve (t½λz) of AZD7503 | 99 days
  To characterise the PK (t½λz) of AZD7503 following SC administration of AZD7503.
Mean residence time of the unchanged drug in the systemic circulation (MRTinf) of AZD7503 | 99 days
  To characterise the PK (MRTinf) of AZD7503 following SC administration of AZD7503.
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) of AZD7503 | 99 days
  To characterise the PK (CL/F) of AZD7503 following SC administration of AZD7503.
Apparent volume of distribution at steady state following extravascular administration based on terminal phase(Vz/F) of AZD7503 | 99 days
  To characterise the PK (Vz/F) of AZD7503 following SC administration of AZD7503.
Time of last observed (quantifiable) concentration (tlast) of AZD7503 | 99 days
  To characterise the PK (tlast) of AZD7503 following SC administration of AZD7503.
Lowest observed drug concentration (Ctrough) before next dose of AZD7503 | 99 days
  To characterise the PK (Ctrough) of AZD7503 following SC administration of AZD7503.
Apparent volume of distribution at steady state following extravascular administration (Vss/F) of AZD7503 | 99 days
  To characterise the PK (Vss/F) of AZD7503 following SC administration of AZD7503.
Accumulation ratio for AUC of AZD7503. | 99 days
  To characterize the PK (Rac AUC) of AZD7503 following SC administration of AZD7503
Accumulation ratio for Cmax (Rac Cmax) of AZD7503 | 99 days
  To characterize the PK (Rac Cmax) of AZD7503 following SC administration of AZD7503.
Partial area under plasma concentration-time-curve from time 0 to time t (AUC(0-t)) of AZD7503 | 99 days
  To characterise the PK (AUC(0-t)) of AZD7503 following SC administration of AZD7503

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: d9230c00003-Redacted_CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9230C00003&attachmentIdentifier=a753d36a-fedb-47e3-ba2c-162fb7879a53&fileName=d9230c00003-Redacted_CSR_synopsis.pdf&versionIdentifier=